CLINICAL TRIAL: NCT02351960
Title: A Phase 4, Open-Label Study in Patients From Asia With Gastroesophageal Reflux Disease Treated With Dexlansoprazole
Brief Title: Dexlansoprazole in Asian Participants With Gastroesophageal Reflux Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEX-P4-001; U1111-1155-8622 (Registry Identifier: WHO)
Record Dates: First submitted 2015-01-27; First posted 2015-01-30 (Estimated); Results first posted 2017-10-04 (Actual); Last update posted 2017-10-04 (Actual); Status verified 2017-05

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Drug therapy; GERD; Dexlansoprazole
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Dexlansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexlansoprazole 30 mg (Experimental): Dexlansoprazole 30 mg, capsules, orally, once daily for up to 4 weeks to participants with non-erosive reflux disease (NERD).
  Interventions: Drug: Dexlansoprazole
- Dexlansoprazole 60 mg (Experimental): Dexlansoprazole 60 mg, capsules orally, once daily for up to 8 weeks to participants with erosive esophagitis (EE).
  Interventions: Drug: Dexlansoprazole

INTERVENTIONS:
Drug: Dexlansoprazole — Dexlansoprazole capsules

SUMMARY:
The purpose of this study is to evaluate the effectiveness of symptom control in gastroesophageal reflux disease (GERD) participants following treatment with dexlansoprazole.

DETAILED DESCRIPTION:
The drug being tested in this study is called dexlansoprazole. A dual delayed release formulation of dexlansoprazole, referred to as dexlansoprazole modified release (dexlansoprazole MR) was tested to treat people who have gastroesophageal reflux disease (GERD). This study looked at the healing of the esophageal lining of the GERD participants who took dexlansoprazole MR.

The study enrolled 296 patients. Participants were assigned to two study groups based on the endoscopy screening procedures to receive treatments as follows:

* Dexlansoprazole 30 mg to participants with non-erosive reflux disease (NERD)
* Dexlansoprazole 60 mg to participants with erosive esophagitis (EE)

All participants were asked to take one capsule in the morning each day throughout the study. All participants were asked to record the presence and maximum severity of daytime and nighttime heartburn and regurgitation symptoms during screening and, if assigned to a treatment group, throughout the duration of the study using the supplied paper diary.

This multi-center trial was conducted in Asia (Hong Kong, Taiwan, South Korea). The overall time to participate in this study was up to 8 weeks. Participants would make up to 3 visits to the clinic, and would be contacted by telephone 30 days after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria: -

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any procedures
3. Has persistent typical gastroesophageal reflux disease (GERD) symptoms (heartburn and/or acid regurgitation) for at least 6 months and a frequency of GERD symptoms is at least 4 days within the past 7 days prior to the screening visit
4. Meets one of the following diagnoses verified by the screening endoscopy

   1. Has macroscopically normal esophageal mucosa on endoscopy and may thereby be eligible for assignment to the nonerosive reflux disease (NERD) study group
   2. Has evidence of erosive esophageal reflux disease on endoscopy, Los Angeles (LA) classification grades B-D, and thereby may be eligible for assignment to the erosive esophagitis (EE) study group
5. Is able and willing to record GERD symptoms in a subject diary and has completed the diary at least for 7 consecutive days during the screening period
6. Male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 30 days after last dose
7. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study
8. All female participants of childbearing potential must have a negative urine pregnancy test at Screening and a negative urine pregnancy test at Day -1. Participants who have had a bilateral tubal ligation, hysterectomy or are post-menopausal (the absence of menses for 1-2 years with a Follicle-Stimulating Hormone [FSH] level >40 IU/L or absence of menses for >2 years) are not required to use birth control

Exclusion Criteria:

1. Has received any investigational compound within 30 days prior to Screening
2. Known hypersensitivity to any proton pump inhibitor (including lansoprazole, omeprazole, rabeprazole, pantoprazole or esomeprazole), any component of dexlansoprazole
3. Use of a H2 blocker or a PPI other than dexlansoprazole during screening and throughout the study. Previous use of Dexlansoprazole before screening
4. Endoscopic Barrett's esophagus and/or definite dysplastic changes in the esophagus
5. Active gastric or duodenal ulcers within 4 weeks of the first dose of study drug
6. History of dilatation of esophageal strictures, other than a Schatzki's ring (a ring of mucosal tissue near the lower esophageal sphincter)
7. Co-existing diseases affecting the esophagus, (eg, esophageal varices, scleroderma, viral, fungal infection or esophageal stricture), history of radiation therapy or cryotherapy to the esophagus, caustic or physiochemical trauma such as sclerotherapy to the esophagus
8. Chronic use (>12 doses/month) of non-;steroidal anti-inflammatory drugs (NSAIDs) including COX 2 NSAIDs within 30 days prior to screening period and throughout the study, however, low dose aspirin up to 325 mg per day is allowed
9. In the judgment of the investigator, participant has clinically significant abnormal hematological parameters of hemoglobin, hematocrit, or erythrocytes at Screening
10. Has a history or clinical manifestations of significant organ failure which would preclude their successful completion of the study
11. Participants using drugs with significant anticholinergic effects such as tricyclics who cannot stay on a stable dose for 4 weeks prior to dosing and throughout the study
12. Participants with known biliary disease
13. Participants with the need for continuous anticoagulant therapy
14. Participants with cancer (except basal cell and squamous cell carcinoma of the skin) within 3 years prior to Screening
15. Any condition that may require inpatient surgery during the course of the study
16. Has abnormal laboratory values that suggest a clinically significant underlying disease or condition that may prevent the subject from entering the study; or subject with the following lab abnormalities: Creatinine >1.5 mg/dL, Alanine Aminotransferase (ALT) and/or Aspartate Aminotransferase (AST) >2.0X the upper limits of normal, or Total Bilirubin >2.0 mg/dL with AST/ALT elevated above normal values
17. Known to have acquired immunodeficiency syndrome (AIDS)
18. Current or historical evidence of Zollinger-Ellison syndrome or other hypersecretory condition
19. History of gastric, duodenal or esophageal surgery except simple oversew of an ulcer
20. Acute upper gastrointestinal (UGI) hemorrhage within 4 weeks of endoscopy

22. Has received blood products within 3 months prior to the first dose of study drug 23. History of alcohol abuse [>21 units (1 unit = 12 oz beer, 1.5 oz hard liquor, or 5 oz wine) per week] or illegal drug use or drug addiction in the 12 months prior to Screening 24. Participants who, in the opinion of the investigator, are unable to comply with the requirements of the study or are unsuitable for any reason 25. is required to take excluded medications 26. If female, the participant is pregnant or lactating or intending to become pregnant before, during, or within 1 month after participating in this study; or intending to donate ova during such time period 27. If male, the participant intends to donate sperm during the course of this study or for 30 days thereafter

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2015-03-19 (Actual); Primary Completion 2016-06-22 (Actual); Study Completion 2016-07-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- Shatin, New Territories, Hong Kong
- South Korea (2):
  - Gyeonggi-do
  - Seoul
- Taiwan (5):
  - Kaoshiung
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan District

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 12 investigative sites in Hong Kong, South Korea, Taiwan from 19 March 2015 to 13 July 2016.
Pre-assignment Details: Participants with a diagnosis of non-erosive reflux disease (NERD) were enrolled to receive dexlansoprazole 30 mg and participants with erosive esophagitis (EE) were enrolled to receive dexlansoprazole 60 mg.
Period: Overall Study
Arm/Group | Dexlansoprazole 30 mg | Dexlansoprazole 60 mg
Started | 208 | 88
Completed | 197 | 76
Not Completed | 11 | 12
Not completed — Pretreatment Event/Adverse Event | 6 | 3
Not completed — Voluntary Withdrawal | 5 | 4
Not completed — Significant Protocol Deviation | 0 | 5

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAF) included all participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexlansoprazole 30 mg | Dexlansoprazole 60 mg | Total
Number analyzed (Participants) | 208 | 88 | 296
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (13.62) | 51.7 (12.51) | 52.6 (13.06)
Age, Customized [Number; unit: participants]
  <45 years | 60 | 29 | 89
  45-<65 years | 102 | 42 | 144
  ≥65 years | 46 | 17 | 63
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 49 | 121
  Male | 136 | 39 | 175
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 208 | 87 | 295
  Multiracial | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Hong Kong | 13 | 6 | 19
  Korea, Republic Of | 195 | 12 | 207
  Taiwan, Province Of China | 0 | 70 | 70
Weight [Mean (Standard Deviation); unit: kg] | 60.26 (11.619) | 68.84 (14.986) | 64.55 (13.302)
Height [Mean (Standard Deviation); unit: cm] | 161.5 (8.43) | 165.0 (9.65) | 163.25 (9.04)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index = weight (kg)/[height (m)^2].
  kg/m^2 | 23.00 (3.305) | 25.11 (4.160) | 24.05 (3.732)
BMI categories [Number; unit: participants]
  <25 kg/m^2 | 158 | 46 | 204
  25-<30 kg/m^2 | 43 | 33 | 76
  ≥30 kg/m^2 | 7 | 9 | 16
Smoking History [Number; unit: participants]
  Never Smoked | 169 | 61 | 230
  Current Smoker | 15 | 11 | 26
  Ex-smoker | 24 | 16 | 40
12-Lead Electrocardiogram (ECG) [Number; unit: participants]
  Within Normal Limits | 141 | 55 | 196
  Abnormal but not Clinically Significant | 67 | 33 | 100

OUTCOME MEASURES:

1. Primary Outcome: Percentage of 24-Hour Heartburn and Acid Regurgitation-Free Days in Non-Erosive Reflux Disease (NERD) Participants
Description: NERD participants were asked to keep a paper diary of daily heartburn and acid regurgitation-free days and the percentage of heartburn and acid regurgitation-free days was recorded.
Time Frame: Up to Week 4
Population: Full analysis set (FAS) included all participants who received at least 1 dose of study drug and had post-baseline data for the appropriate efficacy variable.
Measure: Median (Full Range); unit: percentage of days
Arm/Group | Dexlansoprazole 30 mg
Number analyzed (Participants) | 207
percentage of days | 26.92 [0.0 to 100.0]

2. Primary Outcome: Percentage of 24-Hour Heartburn and Acid Regurgitation-Free Days in Erosive Esophagitis (EE) Participants
Description: EE participants were asked to keep a paper diary of daily heartburn and acid regurgitation-free days and the percentage of heartburn and acid regurgitation-free days was calculated.
Time Frame: Up to Week 8
Population: FAS included all participants who received at least 1 dose of study drug and had post-baseline data for the appropriate efficacy variable. Here number of participants analyzed are the participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: percentage of days
Arm/Group | Dexlansoprazole 60 mg
Number analyzed (Participants) | 87
percentage of days | 65.45 [0.0 to 100.0]

3. Secondary Outcome: Percentage of 24-hour Heartburn-free Days
Description: Participants were asked to keep a daily paper diary. The percentage of 24-hour heartburn free days following study drug treatments was assessed by the participant diary entries.
Time Frame: Up to 4 weeks for NERD participants and up to 8 weeks for EE participants
Population: as for outcome 2
Measure: Median (Full Range); unit: percentage of days
Arm/Group | Dexlansoprazole 30 mg | Dexlansoprazole 60 mg
Number analyzed (Participants) | 207 | 87
percentage of days | 53.85 [0.0 to 100.0] | 81.97 [0.0 to 100.0]

4. Secondary Outcome: Percentage of 24-hour Acid Regurgitation-free Days
Description: Participants were asked to keep a daily paper diary. The percentage of 24-hour acid regurgitation-free days following study drug treatments was assessed by participant's diary entries.
Time Frame: Up to 4 weeks for NERD participants and up to 8 weeks for EE participants
Population: as for outcome 2
Measure: Median (Full Range); unit: percentage of days
Arm/Group | Dexlansoprazole 30 mg | Dexlansoprazole 60 mg
Number analyzed (Participants) | 207 | 88
percentage of days | 75.00 [0.0 to 100.0] | 88.46 [0.0 to 100.0]

5. Secondary Outcome: Percentage of Nights (Participant Sleep Time) Without Nighttime Heartburn and Acid Regurgitation
Description: Participants were asked to keep a daily paper diary. The percentage of nights without nighttime heartburn and acid regurgitation in both the group was assessed by participant dairy entries.
Time Frame: Up to 4 weeks for NERD participants and up to 8 weeks for EE participants
Population: as for outcome 2
Measure: Median (Full Range); unit: percentage of nights
Arm/Group | Dexlansoprazole 30 mg | Dexlansoprazole 60 mg
Number analyzed (Participants) | 207 | 87
percentage of nights | 59.26 [0.0 to 100.0] | 83.33 [0.0 to 100.0]

6. Secondary Outcome: Percentage of Nights (Participant Sleep Time) Without Nighttime Heartburn
Description: Participants were asked to keep a daily paper diary. The percentage of nights without nighttime heartburn in both the group was assessed by participant diary entries.
Time Frame: Up to 4 weeks for NERD participants and up to 8 weeks for EE participants
Population: as for outcome 2
Measure: Median (Full Range); unit: percentage of nights
Arm/Group | Dexlansoprazole 30 mg | Dexlansoprazole 60 mg
Number analyzed (Participants) | 207 | 87
percentage of nights | 73.08 [0.0 to 100.0] | 92.73 [0.0 to 100.0]

7. Secondary Outcome: Percentage of Nights (Participant Sleep Time) Without Nighttime Acid Regurgitation
Description: Participants were asked to keep a daily paper diary. The percentage of nights without nighttime acid regurgitation in both the group was assessed by participant diary entries.
Time Frame: Up to 4 weeks for NERD participants and up to 8 weeks for EE participants
Population: as for outcome 2
Measure: Median (Full Range); unit: percentage of nights
Arm/Group | Dexlansoprazole 30 mg | Dexlansoprazole 60 mg
Number analyzed (Participants) | 207 | 87
percentage of nights | 88.00 [0.0 to 100.0] | 92.59 [0.0 to 100.0]

8. Secondary Outcome: Number of Participants With Severity of Gastroesophageal Reflux Disease (GERD) Symptoms
Description: The severity of participants' GERD symptoms based on the investigator's assessment among all participants was evaluated at Week 4 or Week 8. GERD symptoms were assessed on a 5-point scale, wherein 1=no symptom, 2=mild, 3=moderate, 4=severe and 5=very severe. GERD symptoms include heartburn (HB), acid regurgitation (AR), dysphagia (dysp), belching (bch) and epigastric pain (EP).
Time Frame: Up to 4 weeks for NERD participants and up to 8 weeks for EE participants
Population: FAS included all participants who received at least 1 dose of study drug and had post-baseline data for the appropriate efficacy variable. Here, 'n' is the number of participants who were analyzed for GERD assessments at specified time points.
Measure: Number; unit: participants
Arm/Group | Dexlansoprazole 30 mg | Dexlansoprazole 60 mg
Number analyzed (Participants) | 207 | 88
participants
  Heartburn, None | 77 | 51
  Heartburn, Mild | 92 | 21
  Heartburn, Moderate | 20 | 3
  Heartburn, Severe | 6 | 1
  Heartburn, Very Severe | 3 | 0
  Acid Regurgitation, None | 97 | 52
  Acid Regurgitation, Mild | 76 | 21
  Acid Regurgitation, Moderate | 17 | 3
  Acid Regurgitation, Severe | 7 | 0
  Acid Regurgitation, Very Severe | 1 | 0
  Dysphagia, None | 169 | 71
  Dysphagia, Mild | 22 | 5
  Dysphagia, Moderate | 6 | 0
  Dysphagia, Severe | 1 | 0
  Dysphagi, Very Severe | 0 | 0
  Belching, None | 138 | 57
  Belching, Mild | 46 | 17
  Belching, Moderate | 12 | 2
  Belching, Severe | 1 | 0
  Belching, Very Severe | 1 | 0
  Epigastric Pain, None | 144 | 58
  Epigastric Pain, Mild | 42 | 18
  Epigastric Pain, Moderate | 9 | 0
  Epigastric Pain, Severe | 3 | 0
  Epigastric Pain, Very Severe | 0 | 0

9. Secondary Outcome: Percentage of Participants in the EE Group Who Had Endoscopically Evaluated Macroscopic Healing of Their Esophagus
Description: Participants underwent endoscopy to determine the percentage of participants with macroscopic healing of their esophagus showing at least 1 Los Angeles (LA) grade classification grade improvement at week 8. Endoscopic findings classified according to the Los Angeles classification: Grade Normal - endoscopy reveals no mucosal break Grade A- one or more mucosal breaks <5 mm in maximal length Grade B - one or more mucosal breaks >5 mm, but without continuity across mucosal folds Grade C - Mucosal breaks continuous between >2 mucosal folds, but involving less than 75% of the esophageal circumference Grade D - Mucosal breaks involving more than 75% of the esophageal circumference.
Time Frame: Week 8
Population: FAS included all participants who received at least 1 dose of study drug and had post-baseline data for the appropriate efficacy variable.
Measure: Number; unit: percentage of participants
Arm/Group | Dexlansoprazole 60 mg
Number analyzed (Participants) | 88
percentage of participants | 77.3

ADVERSE EVENTS:
Time Frame: Day 1 up to 30 days after the last dose of study drug (approximately up to 12 weeks)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Dexlansoprazole 30 mg | Dexlansoprazole 60 mg
Serious Adverse Events (participants affected / at risk) | 0/208 | 2/88
Other Adverse Events (participants affected / at risk) | 7/208 | 2/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dexlansoprazole 30 mg (N=208) | Dexlansoprazole 60 mg (N=88)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 — The outcome of the event of adenocarcinoma was fatal and is not related to study drug.
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dexlansoprazole 30 mg (N=208) | Dexlansoprazole 60 mg (N=88)
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Headache (Nervous system disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.